CLINICAL TRIAL: NCT07207460
Title: Comparison of Hydrodissection Techniques Using 5% Dextrose for the Treatment of Carpal Tunnel Syndrome
Brief Title: Hydrodissection in Carpal Tunnel Syndrome
Acronym: KTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Berna Orhan, Physical Therapy and Rehabilitation Specialist, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E2-23-4769
Record Dates: First submitted 2025-09-17; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Carpal Tunnel Syndrome; Median Nerve Entrapment
Keywords: Carpal Tunnel Syndrome; perineural injection; nerve hydrodissection; Conservative treatment; Entrapment neuropathy; 5% dextrose; ultrasound-guided hydrodissection
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy; Charcot-Marie-Tooth Disease | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized, controlled, single-blind trial. Patients diagnosed with mild or moderate CTS based on EMG findings were randomly assigned into three groups using a computerized randomization method. Perineural hydrodissection was performed with 5 mL of 5% dextrose solution in all groups: Group 1 with the in-plane US-guided ulnar approach, Group 2 with the out-of-plane US-guided proximal-to-distal ulnar approach, and Group 3 with the blind proximal-to-distal longitudinal approach. Assessments were conducted at baseline, 2 weeks, and 3 months after the injection. Outcome measures included the Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) and the DN4 questionnaire for CTS severity and functional status, as well as pain intensity assessed using a Visual Analog Scale (VAS). Median nerve cross-sectional area (CSA) was measured at baseline by a physician with over 10 years of US experience, and electromyography (EMG) evaluations were performed at baseline and 3 m
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study was conducted by four independent researchers. One investigator confirmed the CTS diagnosis using EMG and performed all follow-up EMG assessments. A second investigator measured the CSA using ultrasound. A third investigator performed all injections, while a fourth investigator was responsible for clinical evaluations and statistical analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ultrasound-guided in-plane injection technique (Active Comparator): With the patient seated, the lower third of the forearm and the entire palm were sterilized using 2% povidone-iodine. A sterile cover was applied to the ultrasound probe, and sterile gel was placed on the skin. The probe was positioned transversely at the palmar wrist crease at the entrance of the carpal tunnel, allowing visualization of the pisiform, ulnar nerve, and ulnar artery . The ulnar nerve lies just radial to the pisiform, with the ulnar artery located radial to the ulnar nerve; Doppler imaging was used when necessary to confirm arterial position. After identifying the median nerve with ultrasound, a 22-gauge, 38 mm needle was advanced via the ulnar approach. The ulnar nerve and artery were visualized throughout the procedure. The needle was first advanced to the inferior surface of the median nerve with the bevel facing upward; following negative aspiration, 2.5 mL of 5% dextrose solution was injected. Without removing the needle from the skin, the bevel was then r
  Interventions: Procedure: Comparison of three different injection techniques using hydrodissection with 5% dextrose in the treatment of CTS
- ultrasound-guided out-of-plane injection technique (Active Comparator): The patient was seated, and the lower third of the forearm and the entire palm were sterilized with 2% povidone-iodine. A sterile drape covered the ultrasound probe, and sterile gel was applied to the skin. The probe was placed transversely at the proximal wrist crease to visualize the median nerve, then shifted ulnarly to identify the pisiform, ulnar nerve, and ulnar artery. Doppler imaging was used when necessary to confirm arterial position. For the out-of-plane technique, a proximal-to-distal longitudinal approach was employed. With the median nerve visualized, a 22-gauge, 38 mm needle was inserted, and after negative aspiration, 5 mL of 5% dextrose solution was injected between the median nerve and the flexor retinaculum
  Interventions: Procedure: Comparison of three different injection techniques using hydrodissection with 5% dextrose in the treatment of CTS
- blind technique (Active Comparator): This injection technique relies on anatomical landmarks, targeting the space between the palmaris longus tendon and the flexor carpi radialis. The patient was seated, and the lower third of the forearm and the entire palm were sterilized using 2% povidone-iodine. The most commonly used landmarks for the blind approach were the ulnar edge of the palmaris longus tendon and the proximal wrist crease. A 22-gauge, 38 mm needle was inserted at the ulnar border of the palmaris longus tendon along the scaphoid-pisiform line and advanced distally toward the ring finger at an angle of approximately 30°-45°. In patients lacking a palmaris longus tendon, the needle was inserted just ulnar to the wrist midline. Upon patient-reported paresthesia, the needle was slightly withdrawn and redirected ulnarly. Aspiration was performed in all cases to avoid intravascular injection, and 5 mL of 5% dextrose solution was administered slowly and steadily.
  Interventions: Procedure: Comparison of three different injection techniques using hydrodissection with 5% dextrose in the treatment of CTS

INTERVENTIONS:
Procedure: Comparison of three different injection techniques using hydrodissection with 5% dextrose in the treatment of CTS — Comparison of three different injection techniques with D5W
  Other Names: land-mark technique; ultrasound-guided injection technique

SUMMARY:
The aim of this study was to compare the effectiveness of perineural hydrodissection methods performed with 5 mL D5W solution and three different injection techniques [ultrasound-guided in-plane, ultrasound-guided out-of-plane, and blind technique] in cases diagnosed with mild to moderate CTS by EMG.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is a highly prevalent condition in the general population, markedly impairing daily activities and sleep quality. Depending on disease severity and symptom burden, treatment approaches are broadly categorized as conservative or surgical. Beyond lifestyle modifications, numerous conservative interventions-including splinting, extracorporeal shock wave therapy, therapeutic ultrasound, phonophoresis, hydrodissection, kinesiotaping, corticosteroid (CS) injections, low-level laser therapy, platelet-rich plasma (PRP) injections, manual therapy, and acupuncture-have demonstrated clinical efficacy. More recently, 5% dextrose injections have emerged as a safe alternative to CS with minimal adverse effects. Injection therapies vary in both content and technique; however, no consensus exists regarding the optimal approach. Given the importance of minimizing side effects and ensuring long-term effectiveness, the refinement of injection agents and techniques remains a priority. Although ultrasound-guided injections improve safety and accuracy, they require expertise and incur additional costs, whereas blind techniques have long been applied reliably in clinical practice. Nevertheless, comparative studies evaluating these techniques remain limited. Therefore, the present study aimed to compare three different injection techniques for the management of CTS.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 20-70
* Moderate and mild CTS patients diagnosed with CTS by EMG
* Literate patients who agreed to participate in the study

Exclusion Criteria:

* Patients with RA, type 1 or type 2 diabetes mellitus
* Patients with chronic renal failure
* Polyneuropathy
* Those with a history of cancer, those receiving chemotherapy
* Those with a history of broken hand wrist fracture in the last 6 months
* Patients with brachial plexopathy or thoracic outlet syndrome (TOS)
* Patients who underwent surgery due to CTS
* Pregnancy
* Hypothyroidism in a mixed edema picture
* Diagnosed with neuromuscular disease
* Patients with bleeding disorders or those currently receiving anticoagulant therapy
* patients with infection at the injection site

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Boston CTS | 0 , 2nd week 12th week
  The BCTQ is the most widely used measure for CTS. It includes 2 subscales with 11 questions assessing symptom severity and 8 questions assessing functional status.31 Scores range from 0 to 5 points for each question, with higher scores indicating greater severity and dysfunction.The BCTQ provides a standardized, patient-based outcome measure of symptom severity and functional status to assess the results of carpal tunnel syndrome treatments. The test has strong evidence of validity, reliability and responsiveness.
VAS | 0 2nd week 12th week
  VAS was used to assess digital pain intensity and paresthesia/dysthesia before injection therapy administration. Scores ranged from 10 (extremely severe pain) to 0 (no pain).
DN-4 | 0 2nd week 12th week
  It is a clinical screening tool used to diagnose the presence of neuropathic pain.It was developed by the French Neuropathic Pain Group to address the difficulties and lack of consensus in diagnosing neuropathic pain.It is a questionnaire consisting of 10 items administered by the clinician.Seven pain-related items (i.e., sensory and pain descriptors) are administered in consultation with the patient. They express how pain is felt by the patient.The three items are based on clinical examination. The clinician assesses whether sensation to touch or pinprick is diminished (hyposthesia) and whether it increases with light brushing or causes pain (allodynia).

SECONDARY OUTCOMES:
Nerve CSA | 0 2nd 12th week
  The cross-sectional area (CSA) of the median nerve was measured at baseline, 2 weeks, and 3 months after injection by a physician with over 10 years of ultrasound experience. Patients were seated with the forearm supinated and the wrist in slight dorsiflexion, supported by a rolled towel or pillow. A high-frequency linear probe (5-12 MHz, Logic P5, GE Medical Systems) was placed on the palmar wrist in the transverse plane. The median nerve was identified at the level of the scaphoid (radial side) and pisiform (ulnar side), typically in the midline beneath the superficial flexor tendons. CSA was measured by tracing the inner border of the perineural echogenic rim. Each measurement was repeated three times, and the mean value was recorded.
EMG | 0 and 12th week
  Using electrophysiological studies, CTS degree (distal motor latency [DML]) greater than 3.6 was considered as moderate CTS, and those less than 3.6 as mild CTS. Only participants with mild-to-moderate CTS were included in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Berna Orhan, MD, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mathieu T, Lemmens E, Stassijns G. A safe and easy-to-use ultrasound-guided hydrodissection technique for the carpal tunnel syndrome: a minimally invasive approach. J Ultrasound. 2022 Sep;25(3):451-455. doi: 10.1007/s40477-021-00597-5. Epub 2021 Jul 2. PMID 34213741
- [Background] Babaei-Ghazani A, Roomizadeh P, Forogh B, Moeini-Taba SM, Abedini A, Kadkhodaie M, Jahanjoo F, Eftekharsadat B. Ultrasound-Guided Versus Landmark-Guided Local Corticosteroid Injection for Carpal Tunnel Syndrome: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Arch Phys Med Rehabil. 2018 Apr;99(4):766-775. doi: 10.1016/j.apmr.2017.08.484. Epub 2017 Sep 21. PMID 28943161
- [Background] Lee K, Park JM, Yoon SY, Kim MS, Kim YW, Shin JI, Lee SC. Ultrasound-Guided Nerve Hydrodissection for the Management of Carpal Tunnel Syndrome: A Systematic Review and Network Meta-Analysis. Yonsei Med J. 2025 Feb;66(2):111-120. doi: 10.3349/ymj.2024.0089. PMID 39894044
- [Background] Wu YT, Ke MJ, Ho TY, Li TY, Shen YP, Chen LC. Randomized double-blinded clinical trial of 5% dextrose versus triamcinolone injection for carpal tunnel syndrome patients. Ann Neurol. 2018 Oct;84(4):601-610. doi: 10.1002/ana.25332. Epub 2018 Oct 4. PMID 30187524
- [Background] Lee JY, Park Y, Park KD, Lee JK, Lim OK. Effectiveness of ultrasound-guided carpal tunnel injection using in-plane ulnar approach: a prospective, randomized, single-blinded study. Medicine (Baltimore). 2014 Dec;93(29):e350. doi: 10.1097/MD.0000000000000350. PMID 25546691
- [Background] Babaei-Ghazani A, Forogh B, Raissi GR, Ahadi T, Eftekharsadat B, Yousefi N, Rahimi-Dehgolan S, Moradi K. Ultrasound-Guided Corticosteroid Injection in Carpal Tunnel Syndrome: Comparison Between Radial and Ulnar Approaches. J Pain Res. 2020 Jun 26;13:1569-1578. doi: 10.2147/JPR.S248600. eCollection 2020. PMID 32617017
- [Background] Buntragulpoontawee M, Chang KV, Vitoonpong T, Pornjaksawan S, Kitisak K, Saokaew S, Kanchanasurakit S. The Effectiveness and Safety of Commonly Used Injectates for Ultrasound-Guided Hydrodissection Treatment of Peripheral Nerve Entrapment Syndromes: A Systematic Review. Front Pharmacol. 2021 Mar 5;11:621150. doi: 10.3389/fphar.2020.621150. eCollection 2020. PMID 33746745
- [Background] Cage ES, Beyer JJ, Ebraheim NA. Injections for treatment of carpal tunnel syndrome: A narrative review of the literature. J Orthop. 2023 Feb 21;37:81-85. doi: 10.1016/j.jor.2023.02.011. eCollection 2023 Mar. PMID 36974095
- [Background] Borire AA, Hughes AR, Lueck CJ, Colebatch JG, Krishnan AV. Sonographic differences in carpal tunnel syndrome with normal and abnormal nerve conduction studies. J Clin Neurosci. 2016 Dec;34:77-80. doi: 10.1016/j.jocn.2016.05.024. Epub 2016 Jul 25. PMID 27469410